CLINICAL TRIAL: NCT03197246
Title: May Intravascular Electrocardiography (IVECG) During Insertion of Peripheral Inserted Central-venous Catheters (PICC-line) Replace Chest X-ray?
Brief Title: Intravascular ECG During Insertion of Peripheral Inserted Central-venous Catheters: Replacement for Chest X-ray?
Acronym: IVEKG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SPL4911
Record Dates: First submitted 2017-06-15; First posted 2017-06-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Catheterization, Peripheral; Electrocardiography
Keywords: PICC line; ECG; chest x-ray; IVECG; ICECG
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Intervention Model Description: RCT, two groups
Who Masked: Outcomes Assessor
Masking Description: The radiologist is masked/blinded in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVECG and chest X-ray (Experimental): The patients in this group will be examined with perioperative IVECG for PICC tip placement, as well as standard postoperative chest X-ray.
  Interventions: Device: IVECG; Device: Chest X-ray
- Standard (Active Comparator): Standard method, PICC tip placement confirmed by postoperative chest X-ray .
  Interventions: Device: Chest X-ray

INTERVENTIONS:
Device: IVECG — Monitoring IVECG signals for verification for exact tip placement during the actual insertion of the PICC. When the p-wave amplitude increases the PICC-tip is in the superior vena cava. When max positive amplitude, the PICC-tip is by definition at the cavo atriale junction, and thereby in correct position.
  Other Names: intravascular electrocardiography
  Arms: IVECG and chest X-ray
Device: Chest X-ray — Standard method; PICC confirmed by chest X-ray after the insertion (postoperatively)

SUMMARY:
This study will provide further knowledge concerning the use of electrocardiography (ECG) signals for verification of peripherally inserted central catheter (PICC) tip placement. Furthermore, it will be investigating whether use of Intravascular ECG (IVECG) for this verification is just as good as or even better than the current standard method with chest X-ray. This can help promote a method that involves less radiation and increased safety for patients, while at the same time saving resources. If use of ECG signals from the PICC tip is an equally exact method for verification of correct PICC tip placement as chest X-ray verification, the IVECG could replace chest X-ray control.

ELIGIBILITY:
Inclusion Criteria:

* In need for PICC
* >18 years old
* Competent to give consent

Exclusion Criteria:

* Not visible p-wave on surface ECG (electrocardiograph)
* Patients with known Atrial fibrillation or atrial flutter
* Implanted pacemaker (PM) and/or implanted Implantable Cardioverter Defibrillator (ICD)
* Not signed written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
PICC-tip placement examined by chest X-ray | 45 minutes
  Placement of PICC-tip examined by chest X-ray both in observation group and in control group. A radiologist will examine the distance from the tracheal carina to the PICC-tip, and this measure will be registered in mm in both groups. Further the radiologist will be answering a questionnaire regarding "correct placement of PICC-tip", YES or NO, which is defined as in the lower 1/3 of the superior vena cava or at the cavo atrial junction. Last also the anesthesiologist will be answering following question: Is the PICC-tip placement acceptable? YES or NO

CONTACTS AND LOCATIONS:
Overall Officials: Baard Olav Jensen, MD,PhD, Study Chair — Sykehuset Innlandet HF; Jon Magnussen, prof, Study Director — NTNU, MH, Masterutdanning
Locations (1):
- Innlandet Hospital Trust Lillehammer, Lillehammer, Oppland, Norway

IPD SHARING:
Plan to Share IPD: No
This is a small project that will not produce any large amount of data. Thus, sharing data for other projects than described to the ethical committee is not relevant. So this is not the plan at this moment.